CLINICAL TRIAL: NCT06940973
Title: Prospective Observational Study of the Morphokinetics and Ploidy of Blastocysts With Abnormal Fertilization (1PN, 2.1PN and 3PN) to Identify the Origin of Fertilization Alterations
Brief Title: Study of Abnormally Fertilized Embryos
Acronym: SAFE
Status: Not yet recruiting | Type: Observational
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: EJC-SAFE-24-02
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Infertility (IVF Patients)
Keywords: PGT-A; niPGT-A; Blastocyst; Infertility; In vitro fertilization; Ploidy; Embryo development; Time-lapse culture; Triploid; Haploid; Abnormal fertilization; Pronuclei
MeSH Terms: conditions — Infertility; Triploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cummulus cells and seminal plasma or saliva from both parents. Blastocyst trophectoderm biopies. Spent blastocyst media with embryonic cell-free DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blastocysts from abnormally fertilized oocytes during assisted reproduction: During the conventional ICSI/IVF procedures in the laboratory, the embryologist observing fertilization will identify embryos with an abnormal pronuclear pattern and preselect them for the study. These embryos will be cultured in a time-lapse incubator following the laboratory's standard practice. All recorded morphokinetic parameters, along with the corresponding images, will be documented. Each embryo will be monitored, its developmental quality assessed and recorded to determine whether it reaches the blastocyst stage. If so, the researchers will contact the patient to ask consent for these embryos to be included in the study.
  Embryos with an abnormal pronuclear pattern that fail to reach the blastocyst stage due to developmental blockage will be discarded.
  No drugs or medical devices will be used.
  Interventions: Genetic: Parental samples; Diagnostic Test: PGT-A; Genetic: TE rebiopsies and spent blastocyst media collection

INTERVENTIONS:
Genetic: Parental samples — On fertilization, following the conventional ICSI/IVF procedure, samples from cumulus cells (obtained during the routine oocyte denudation process) and surplus sperm cells present in seminal plasma will be retrieved. These samples will be stored frozen at -20°C until they are sent to Igenomix. There, they will be used to perform the genetic analysis required to achieve the study's objectives, provided the patient consents to participate. If the patient ultimately chooses not to participate, these samples will be destroyed.
  Parents may be asked to provide a saliva sample for the same purpose in cases where obtaining the samples during fertilization was not possible or if the collected samples were unsuitable for processing in the laboratory. The saliva sample may be collected at the clinic during one of the scheduled visits for reproductive treatment or, alternatively, by the parents at home using a kit provided by the clinic.
Diagnostic Test: PGT-A — On day 3 of development, assisted hatching will be performed to facilitate biopsy at the blastocyst stage. Each embryo will be biopsied in the laboratory using conventional trophectoderm (TE) biopsy techniques on day +5, +6, or +7 of development, depending on when they reach the appropriate blastocyst stage. After biopsy, blastocyst will be vitrified following the clinical routine protocol and store until the genetic results are available. The biopsy samples will be placed in a PCR tube labeled with its corresponding study-specific code and stored in a cold rack at 4°C before being transferred to a freezer at -20°C. Finally, the samples will be sent to the Igenomix for preimplantation genetic testing for aneuploidy.
Genetic: TE rebiopsies and spent blastocyst media collection — After obtaining the PGT-A results, any embryo not genetically confirmed as euploid and without ploidy abnormalities will be thawed, washed, and cultured for rebiopsy. A complementary analysis using next-generation sequencing (NGS) techniques will be performed to confirm the diagnosis and determine the origin of the abnormalities. For this additional analysis, in addition to the new biopsies, the individual culture medium of each embryo will be aspirated after an incubation period of 8 to 24 hours. The collected medium will be placed in PCR tubes and stored in a freezer at -20°C before being sent to the laboratory.
  Regardless the result of these complementary analysis, no rebiopsied blastocyst will be considered for clinical purposes.

SUMMARY:
The goal of this observational study is to determine the diploidy rate of haploid and triploid embryos from in vitro fertilization (IVF) cycles. The main questions it aims to answer are:

* Can a molecular genetic fertilization check of abnormally fertilized embryos be used to expand opportunities for couples undergoing assisted reproduction treatment?
* Is the chromosomal loss or gain present in abnormally fertilized embryos predominantly maternal in origin?

For this purpose, we will evaluate the morphokinetics and ploidy of about 300 embryos with different types of abnormal pronuclear patterns (1PN, 2.1PN, and 3PN) that reach the blastocyst stage. Whenever possible, embryos with a non-diploid chromosomal complement will also be assessed to determine the origin (maternal or paternal) of the chromosomal set that has been lost or gained.

Study subjects will follow their previously scheduIed IVF/ICSI treatment and no additional visits/interventions will be required for participating.

DETAILED DESCRIPTION:
Chromosomes are cellular structures containing the majority of the genetic information of a living organism. Gametes (oocytes and spermatozoa) contain only a single set of 23 chromosomes within structures known as pronuclei (PN). Upon fertilization, the 23 chromosomes from the oocyte and the 23 chromosomes from the sperm combine to form a 2PN zygote, which contains a total of 46 chromosomes.

In assisted reproduction (ART) laboratories, the embryologists can determine through morphological evaluation whether the fertilization process was normal (2PN) or abnormal (0PN, 1PN, or >2PN). For an ART treatment, only a successfully fertilized oocyte (2PN) that develops to the blastocyst stage may be suitable for embryo transfer. However, previous studies have demonstrated that some embryos from oocytes with abnormal fertilization may possess a normal chromosomal content and could be used in ARTs when embryos from normal fertilization are not available.

There are genetic analysis techniques to determine not only if an embryo is euploid (contains a normal number of chromosomes) but also to assess if it is haploid, diploid or triploid (1PN, 2.1PN, and 3PN respectively). These techniques may be applied to "rescue" embryos with abnormal fertilization that are currently being discarded. This approach could be beneficial for IVF patients with a limited number of viable embryos available (diminished ovarian reserve cases, advanced maternal age, poor response to ovarian stimulation, etc.).

The current prospective and observational study has been approved by the competent Research Ethics Committee and every potential participant will be asked to sign the study informed consent.

The 300 embryos that will be part of the study will be recruited in the laboratory of the collaborating center on the day of fertilization after performing the conventional IVF procedures. Following these same routine procedures, biological samples from both parents will also be stored to perform the genetic analysis to determine the origin of the chromosomal anomalies. A biopsy will be taken from the selected embryos when they reach the blastocyst stage for the genetic analysis that will allow detecting whether there is indeed any chromosomal anomaly. All embryos not confirmed as chromosomally normal will be thawed, washed, and cultured for a second biopsy to confirm their previous diagnosis and the origin of the chromosomal abnormalities. For this new analysis, in addition to the biopsies, individual samples of the culture media of the thawed blastocysts will be collected and stored. Samples will be shipped to Igenomix for the genetic research and further data analysis.

The expected duration of the study is 18 months. Embryos will be included in the participating center for an estimated period of 13 months. Participants involvement in the study is just linked to the moment of the consent form signature. Exceptionally, embryos from abnormal fertilization that were informed as chromosomally normal after the first biopsy can be considered to transfer providing there are no other embryos available. If the patient decides to proceed with the transfer, her clinical follow-up will be part of the study until achieving ongoing pregnancy (12 gestational weeks). After that, her participation in the study will end but her physician will continue monitoring the pregnancy until delivery, if applicable, in accordance with the standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* ART patients who sign the Informed Consent of the study.
* Age: oocytes from women ≤ 49 years and semen from men ≤ 60 years. Donation of gametes is allowed.
* ≥1 blastocysts from oocytes with an abnormal pronuclear pattern (1PN, 2.1PN, and/or 3PN) and with the presence of 2 polar bodies (PB), cultured in a time-lapse incubator.

Exclusion Criteria:

* No exclusion criteria have been considered for this study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Embryos from subjects undergoing assisted reproductive treatment with oocytes exhibiting an abnormal number of pronuclei (1PN, 2.1PN, and/or 3PN). Recruitment of subjects for the study will be conducted through routine consultation with the principal investigator and collaborators, as long as they meet the selection criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Diploidy rate in haploid embryos from IVF/ICSI | 3 months
  Number of 2PN blastocysts from abnormally fertilized oocytes (1PN)
Diploidy rate in triploid embryos from IVF/ICSI | 3 months
  Number of 2PN blastocysts from abnormally fertilized oocytes (2.1PN and 3PN)

SECONDARY OUTCOMES:
Origin of the chromosomal abnormalities in embryos with a non-diploid chromosomal content | 6 months
  To determine the origin (maternal or paternal) of the chromosomal set that has been lost or gained.
Pregnancy rate of euploid embryos from abnormal fertilization | 2 weeks after the embryo transfer
  Number of patients with positive serum level of β-human chorionic gonadotropin (βhCG > 25 mIU/ml) per embryo transfer. Beta-hCG will be measured at day 12±2 after the embryo transfer.
Implantation rate of euploid embryos from abnormal fertilization | Up to 4 weeks after the embryo transfer
  Number of gestational sacs observed by vaginal ultrasound divided by the number of embryos transferred.
Biochemical pregnancy rate of euploid embryos from abnormal fertilization | 4 weeks after the embryo transfer with euploid embryos from abnormal fertilization
  Number of pregnancies diagnosed only by β-hCG detection without a gestational sac visualized by vaginal ultrasound, per number of pregnancies.
Ectopic pregnancy rate of euploid embryos from abnormal fertilization | 4-5 weeks after the embryo transfer
  Number of pregnancies outside the uterine cavity, diagnosed by ultrasound, surgical visualization or histopathology, per number of pregnancies.
Clinical miscarriage rate of euploid embryos from abnormal fertilization | Up to 12 gestational weeks
  Number of spontaneous pregnancy losses before week 12, in which a gestational sac/s was previously observed, per number of pregnancies.
Ongoing pregnancy rate of euploid embryos from abnormal fertilization | Over 12 gestational weeks
  Number of pregnancies up to 12 gestational weeks (at least one fetus with a discernible heartbeat diagnosed) achieved per each embryo transfer.
Voluntary termination rate of euploid embryos from abnormal fertilization | Up to 12 gestational weeks
  Number of voluntary terminations before week 12 per number of pregnancies.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Mir Pardo, PhD, Principal Investigator — Igenomix; Carmen Rubio Lluesa, PhD, Principal Investigator — Igenomix
Locations (1):
- Equipo Médico Crespo Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided